CLINICAL TRIAL: NCT00277758
Title: A Phase I Study of Low Dose Interleukin 2 (IL-2)Monotherapy, Followed by IL-2 Plus PEG-IFN/RBV In Chronic Hepatitis C Virus Genotype I Infection
Brief Title: Safety Study of Low Dose Interleukin 2 (IL-2) Plus PEG-IFN/RBV In Chronic Hepatitis C Virus Genotype I
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient rate of volunteer accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Kendall A. Smith, Professor of Medicine, weill Medical College of Cornell University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-092; U01AI048224 (NIH)
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Hepatitis C
Keywords: Interleukin-2
MeSH Terms: conditions — Hepatitis C | interventions — Interleukin-2; aldesleukin; Ribavirin; peginterferon alfa-2b; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Interventions: 12 weeks of interleukin-2 administration, followed by 48 weeks of interleukin-2 + Ribavirin + interferon-alpha therapy, followed by 24 weeks off therapy
  Interventions: Biological: Interleukin 2; Drug: Ribavirin; Biological: Pegylated Interferon Alpha; Biological: Inteleukin-2
- 2 (Active Comparator): 48 weeks of therapy with Ribavirin + interferon-alpha, followed by 24 weeks off therapy
  Interventions: Drug: Ribavirin; Biological: Pegylated Interferon Alpha; Drug: Ribavirin + Pegylated interferon-alpha

INTERVENTIONS:
Biological: Interleukin 2 — Interleukin-2 at 1.2 mU/M2 administered subcutaneously daily
  Other Names: Proleukin
  Arms: 1
Drug: Ribavirin — Ribavirin @ 800 mg daily (< 65 kg body weight), 1000 mg (65-85 kg), and 1200 mg (> 85 kg)
  Other Names: Rebetrol
Biological: Pegylated Interferon Alpha — Pegylated-Interferon-alpha 1.5 ug/kg weekly subcutaneously.
  Other Names: PEG-Intron
Biological: Inteleukin-2 — Interleukin-2 administered as a daily subcutaneous injection at 1.2 mU/M2 BSA
  Other Names: Ribavirin; Interferon-alpha
  Arms: 1
Drug: Ribavirin + Pegylated interferon-alpha — Pegylated interferon-alpha administered 1.5 ug/kg weekly. Ribivirin 800 mg daily for body weight <65 kg, 1000 mg for body weight 65-85 kg, and 1200 mg for body weight >85 kg.
  Other Names: PEG-Intron; Rebetrol
  Arms: 2

SUMMARY:
This is a treatment study trial, in which we will assess the safety and tolerability of daily dose IL-2, as monotherapy for 12 weeks, followed by IL2 in combination with PEG-IFN and RBV for 48 weeks in the treatment of chronic Hepatitis C.

DETAILED DESCRIPTION:
This is a single center study of 12 weeks of IL-2 lead in immunotherapy followed by 48 weeks of IL2 immunotherapy in combination with Pegylated Interferon Alpha (PEG-IFN-alpha) /Ribavirin (RBV) antiviral therapy for the treatment of individuals infected with Hepatitis C virus (HCV) genotype I. The study is designed to determine whether immunotherapy immunotherapy with low dose daily IL-2 can be safely added to the standard antiviral therapy of 48 weeks of PEG-IFN and RBV. Because IL-2 targets recently antigen- activated T cells, IL-2 therapy will be initiated 12 weeks before PEG-IFN/RBV therapy, when HCV antigen load is high, to activate and expand HCV antigen-specific T cells prior to the initiation of antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age >18 years to < 65 years.
* Ability and willingness to sign an informed consent.
* Hepatitis C antibody positive status confirmed by the NYPH laboratory.
* Genotype 1 HCV confirmed by the NYPH laboratory using the DupliType assay as performed by Quest Diagnostics.
* Liver biopsy demonstrating chronic hepatitis but without cirrhosis within 2 years of enrollment.
* Prothrombin time < 3 seconds longer than control.
* Platelet count ≥75,000 mm3
* Neutrophil count ≥ 1000/mm3
* Hemoglobin ≥12 g/dL for women and ≥13 g/dL for men
* Subject must agree not to participate in a conception process (defined as active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization etc.) while on study drugs and for 6 months following permanent discontinuation of study therapy.

Women of reproductive potential (defined for this study as sexually mature women who have not been post-menopausal for at least 24 consecutive months, or have not undergone hysterectomy or oophorectomy) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 MIU/mL performed within 30 days prior to enrollment and again within 24 hours before initiating study therapy.

All subjects must not participate in a conception process, and if participating in sexual activity that could lead to pregnancy, male subjects must take every precaution to avoid risk of pregnancy for their female partners, women subjects/male partners must use two reliable methods of contraception simultaneously, while receiving study therapy and for 6 months following permanent discontinuation of study therapy.

NOTE A: Reliable forms of contraception are a combination of two of the following methods: 1) condoms (male or female) with or without a spermicidal agent. 2) diaphragm or cervical cap with spermicide, 3) IUD, or 4) hormonal-based contraception.

NOTE B: An IUD is an adequate method of contraception but increases the risk of pelvic inflammatory disease.

Exclusion Criteria:

* Previous IFN-alpha, RBV or IL2 therapy
* Any active viral hepatitis other than hepatitis C virus infection, as defined by the presence of IgM antibody to Hepatitis A Virus (HAV) within 30 days of enrollment, or Hepatitis B Virus Surface Antigen (HBsAg) positivity, or positive plasma HBV DNA by PCR methodology when HB core antibody is the only serologic marker of HBV infection within 30 days of entry.
* ALT and AST > 5x ULN, total bilirubin > 1.5 x ULN
* Signs/symptoms of advanced liver disease.
* Uncontrolled infection, except hepatitis C
* HIV infection as determined by HIV ELISA & Western blot assay, and confirmed by plasma HIV assay (PCR or bDNA)
* Cardiac condition that cannot be controlled by medication: Because of the risk of anemia associated with RBV use and the potential to induce cardiac ischemia, subjects with a positive cardiac stress test are ineligible. Therefore, subjects > 40 years of age with ≥ 1 risk factor for ASHD (i.e., hyperlipidemia, hypertension, smoking history, family history) should have an EKG preformed. If the EKG is abnormal and consistent with ischemic heart disease, the subject should have a cardiac stress test to R/O ASHD.
* CNS or psychiatric illness uncontrolled by medication. In particular, psychiatric illness, especially depression. Subjects with a psychiatric illness, a previous suicide attempt or hospitalization for a psychiatric Dx Will be enrolled at the discretion of the investigator.
* Concurrent therapy with any immune-modulating agents, e.g,. interleukins, interferons, therapeutic vaccines, corticosteroids, immunosuppressive agents (azathioprine, 6-mercaptopurine, Cyclosporine-A, FK506, Rapamycin, antilymphocyte antibodies).
* Pregnant or nursing women (all women of child bearing age should be using effective contraception)
* History of malignancy with receipt of cancer therapy within 24 weeks.
* Any severe illness that would make the subject unsuitable for the study.
* Active asthma, or asthma uncontrolled by medication.
* Any immunologically mediated disease, including Crohn's disease, ulcerative colitis, rheumatoid arthritis, lupus erythematosis, ITP, autoimmune hemolytic anemia, eczema, psoriasis.
* Untreated thyroid disease.
* Heroin or cocaine use within 9 months of enrollment.
* Inadequate venous access.

NOTE: If screening TSH is abnormal, obtain free thyroxin index. If the free thyroxine index is normal, the subject may enter the study. If the free thyroxin index is low, the subject may be treated with thyroid hormone replacement medication and enter the study once the free thyroxin index is corrected. If the free thyroxin index is elevated indicating hyperthyroidism, the subject should not enroll in the study.

Patients with preexistent antibodies against thyroid peroxidase or thyroglobulin should not be enrolled.

* Allergy to any of the medications to be used in the study (i.e., IL2, PEG-IFN/RBV), or other components of the study products. Peg Intron: benzyl alcohol, NaCl, Na-phosphate, EDTA, polysorbate 80, m-cresol, IL2; phosphate buffer, SDS, mannitol. RBV: cellulose, lactose, croscarmellose, magnesium stearate, Blue pharmaceutical ink: shellac, anhydrous ethyl alcohol, isopropyl alcohol, n-butyl alcohol, propylene glycol, ammonium hydroxide, Blue # 2 aluminum lake.
* Alcohol dependency, for example, current alcohol use of more than 1 drink/day any time during the previous 6 months. One drink is defined as 12 ounces of beer, 5 ounces of wine, or 1-¼ ounces of hard liquor.
* Severe retinopathy due to diabetes, hypertension, CMV, or macular degeneration
* Acute therapy for a serious infection or other serious medical illness that is potentially life threatening and requires systemic therapy and/or hospitalization within 14 days of study entry.
* Serum creatinine > 2.0 mg/dL or creatinine clearance < 50 mL/min as estimated by the Cockcroft-Gault equation. This screening value must be obtained within 30 days of enrollment.
* History of major organ transplantation with an existing graft.
* Subject judged by the investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results.
* Subjects with biopsy proven liver disease other than HCV infection.
* Subjects with hemoglobinopathies or any other causes or tendencies toward hemolysis.
* Subjects with chronic pulmonary disease with functional limitations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-03; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Determination of the safety and tolerability of 12 weeks IL2 monotherapy followed by 48 weeks of IL2 combined with PEG-IFN/RBV | 60 weeks of therapy followed by 24 weeks off therapy

SECONDARY OUTCOMES:
Determination of specific immunologic responses to HCV. Immunologic assessment will be performed as the sme time intervals as the assays for plasma virus. | 60 weeks of therapy followed by 24 weeks off therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kendall A Smith, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States